CLINICAL TRIAL: NCT06466200
Title: Validation of a French Version of the DHEQ - Oral Health-related Quality of Life and Dentin Hypersensitivity
Brief Title: Validation of a French Version of the DHEQ
Acronym: DHEQ-VALID
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RBHP 2024 DOMEJEAN; 2024-A00861-66 (Other: ANSM)
Record Dates: First submitted 2024-06-11; First posted 2024-06-20 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Dentin Hypersensitivity; Quality of Life
Keywords: Oral health; Dentin Hypersensitivity; Quality of Life
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Intervention Model Description: During their management in the 3 study centers, if the diagnosis of dentin hypersensitivity (DH) is made, a patient may be offered to participate in the study. The group of patients without DH (control group) will consist of patients who meet the inclusion and non-inclusion criteria and who agree to participate.
  Participants will answer the questionnaires on their first visit. A second visit will be organized for the 60 patients randomly selected for a re-test at 15 days.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dentin hypersensitivity group (Other): patients with at least one tooth with a diagnosis of dentin hypersensitivity (DH) with dentin exposure related to gum recession and/or erosive lesion or with a diagnosis of DH with a gingival margin flush with the amelocementary junction. In patients with multiple teeth with DH, the study will consider the most painful tooth according to the EVA score on the air jet test.
  Interventions: Diagnostic Test: Schiff Test; Other: GOHAI questionnaire; Other: OHIP questionnaire; Other: DHEQ fr questionnaire
- control group (Other): Control group: The group of patients without DH will consist of patients from the study centers who meet the inclusion criteria and agree to participate.
  Interventions: Diagnostic Test: Schiff Test; Other: GOHAI questionnaire; Other: OHIP questionnaire; Other: DHEQ fr questionnaire

INTERVENTIONS:
Diagnostic Test: Schiff Test — Use of an air syringe positioned perpendicular to the tooth surface at a distance of 1 cm. A scale to determine the intensity of DH was created, with the SASS (Shiff Analog Sensitivity Scale) ranging from 0 to 3 (0 being the absence of pain felt by the patient and 3 being pain considered intolerable). If the pain is greater than 1 then the patient is considered hypersensitive.
Other: GOHAI questionnaire — Oral health-related quality of life assessment by questionnaire
Other: OHIP questionnaire — Oral health-related quality of life assessment by questionnaire
Other: DHEQ fr questionnaire — dentin hypersensitivity and oral health-related quality of life assessment by questionnaire

SUMMARY:
Dentin hypersensitivity (DH) results in brief, sharp pain in response to a stimulus. It often seems to be underdiagnosed but also undertreated due to the lack of consensus on the topic. DH has been shown to affects patients' quality of life. The Dentine Hypersensitivity Experience Questionnaire (DHEQ)is developed and validated : which is questionnaire assessing specifically the impact of DH on patient's quality of life. The DHEQ aims to help diagnose DH and assess the impact and subjective experience of the patient in order to better meet their expectations in terms of treatment. A French version, the DHEQ-fr, has been proposed (translation-counter-translation process and pilot study); however, it has not yet been validated (psychometric tests, test-retest).

The main objective of the present study is to validate DHEQ-fr through a multicenter clinical study (three centers in France) in adult patients. The secondary objective is to compare the results of DHEQ-fr with those of the general oral health assessment index and oral health impact profil for the same patients. Patients are split between three DH groups (Schiff scores 1, 2 and 3) and a control group (non-DH). The overall sample size (all centers considered) for the DH group is 162 subjects divided into 54 subjects for each Schiff score (1 to 3; after cold air stimulation), with a control group of 54 subjects. A re-test will be performed, at 15 days, on a random sample of 60 subjects from the study population (in total: 15 non-DH subjects; 15 with a Schiff score of 1; 15 with a score of 2; 15 with a score of 3). The study of psychometric properties such as acceptability, internal consistency, reproducibility and internal structure validity will allow the validation of this French version of the DHEQ.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are able to understand the study

Exclusion Criteria:

* Teeth with other pathologies in addition to HD (carious lesions, cracked enamel, etc.);
* Abutment teeth for fixed or removable dentures and crown teeth;
* Teeth with restorations involving the inner third of the dentin and/or restorations involving the dentinary/root exposure area;
* Patients who have been on or have undergone desensitizing therapy for HD in the past three months;
* Patients who have received periodontal surgery within the last three months;
* Patients with orthodontic devices who have interrupted orthodontic treatment in the last three months;
* Pregnant or breastfeeding patients;
* Patients under guardianship, curatorship, safeguard of justice
* Patients deprived of liberty
* Patients participating in any other clinical study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2024-06-25 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
the DHEQ-fr questionnaire | one year
  The 50 items constituting the original questionnaire can be divided in the following sections :
  Items #1-6: description of the sensations related to the pathology Items #7-9: scoring, using a visual analogue scale (VAS), of the intensity, the bothersomeness and the tolerability related to DH Items #10-45: scoring, using a seven-point Likert scale, of the impact of DH on QoL. Five domains or impact subscales can be identified: functional restriction (five items), adaptation (12 items), social impact (five items), emotional impact (eight items) and identity (six items) Item #46: A global oral health rating, with responses on a five-point Likert scale (from "excellent" to "very poor") Items #47-50: The questionnaire also contains four items recording the impact of the sensations on life overall, with responses on a five-point Likert scale (from "not at all" to "very much")

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Domejean, Principal Investigator — CHU de Clermont-Ferrand
Locations (3):
- France (3):
  - CHU de Bordeaux, Bordeaux
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - Centre de soins bucco-dentaires, Lyon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Canadian Advisory Board on Dentin Hypersensitivity. Consensus-based recommendations for the diagnosis and management of dentin hypersensitivity. J Can Dent Assoc. 2003 Apr;69(4):221-6. PMID 12662460
- [Background] West NX, Sanz M, Lussi A, Bartlett D, Bouchard P, Bourgeois D. Prevalence of dentine hypersensitivity and study of associated factors: a European population-based cross-sectional study. J Dent. 2013 Oct;41(10):841-51. doi: 10.1016/j.jdent.2013.07.017. Epub 2013 Aug 1. PMID 23911597
- [Background] Favaro Zeola L, Soares PV, Cunha-Cruz J. Prevalence of dentin hypersensitivity: Systematic review and meta-analysis. J Dent. 2019 Feb;81:1-6. doi: 10.1016/j.jdent.2018.12.015. Epub 2019 Jan 11. PMID 30639724
- [Background] Martinez-Ricarte J, Faus-Matoses V, Faus-Llacer VJ, Flichy-Fernandez AJ, Mateos-Moreno B. Dentinal sensitivity: concept and methodology for its objective evaluation. Med Oral Patol Oral Cir Bucal. 2008 Mar 1;13(3):E201-6. PMID 18305444
- [Background] Holland GR, Narhi MN, Addy M, Gangarosa L, Orchardson R. Guidelines for the design and conduct of clinical trials on dentine hypersensitivity. J Clin Periodontol. 1997 Nov;24(11):808-13. doi: 10.1111/j.1600-051x.1997.tb01194.x. PMID 9402502
- [Background] Schiff T, Dotson M, Cohen S, De Vizio W, McCool J, Volpe A. Efficacy of a dentifrice containing potassium nitrate, soluble pyrophosphate, PVM/MA copolymer, and sodium fluoride on dentinal hypersensitivity: a twelve-week clinical study. J Clin Dent. 1994;5 Spec No:87-92. PMID 8534380
- [Background] Bekes K, John MT, Schaller HG, Hirsch C. Oral health-related quality of life in patients seeking care for dentin hypersensitivity. J Oral Rehabil. 2009 Jan;36(1):45-51. doi: 10.1111/j.1365-2842.2008.01901.x. PMID 19207369
- [Background] Atchison KA, Dolan TA. Development of the Geriatric Oral Health Assessment Index. J Dent Educ. 1990 Nov;54(11):680-7. PMID 2229624
- [Background] Slade GD, Spencer AJ. Development and evaluation of the Oral Health Impact Profile. Community Dent Health. 1994 Mar;11(1):3-11. PMID 8193981
- [Background] Wong AH, Cheung CS, McGrath C. Developing a short form of Oral Health Impact Profile (OHIP) for dental aesthetics: OHIP-aesthetic. Community Dent Oral Epidemiol. 2007 Feb;35(1):64-72. doi: 10.1111/j.1600-0528.2007.00330.x. PMID 17244139
- [Background] McGrath C, Wong AH, Lo EC, Cheung CS. The sensitivity and responsiveness of an oral health related quality of life measure to tooth whitening. J Dent. 2005 Sep;33(8):697-702. doi: 10.1016/j.jdent.2005.01.012. Epub 2005 Mar 19. PMID 16139701
- [Background] Boiko OV, Baker SR, Gibson BJ, Locker D, Sufi F, Barlow AP, Robinson PG. Construction and validation of the quality of life measure for dentine hypersensitivity (DHEQ). J Clin Periodontol. 2010 Nov;37(11):973-80. doi: 10.1111/j.1600-051X.2010.01618.x. Epub 2010 Sep 22. PMID 20860720
- [Background] Machuca C, Baker SR, Sufi F, Mason S, Barlow A, Robinson PG. Derivation of a short form of the Dentine Hypersensitivity Experience Questionnaire. J Clin Periodontol. 2014 Jan;41(1):46-51. doi: 10.1111/jcpe.12175. Epub 2013 Nov 19. PMID 24117603
- [Background] He SL, Wang JH, Wang MH. Development of the Chinese version of the Dentine Hypersensitivity Experience Questionnaire. Eur J Oral Sci. 2012 Jun;120(3):218-23. doi: 10.1111/j.1600-0722.2012.00962.x. PMID 22607338
- [Background] He SL, Wang JH. Reliability and validity of the Chinese version of the short form of the Dentine Hypersensitivity Experience Questionnaire (DHEQ-15). Qual Life Res. 2015 Jun;24(6):1465-9. doi: 10.1007/s11136-014-0856-8. Epub 2014 Nov 9. PMID 25381644
- [Background] Basaran S, Celik C. Turkish Adaptation of Dentine Hypersensitivity Experience Questionnaire (DHEQ). Community Dent Health. 2018 Mar 1;35(1):47-51. doi: 10.1922/CDH_4151Basaran05. PMID 29369544
- [Background] Douglas-De-Oliveira DW, Lages FS, Paiva SM, Cromley JG, Robinson PG, Cota LOM. Cross-cultural adaptation of the Brazilian version of the Dentine Hypersensitivity Experience Questionnaire (DHEQ-15). Braz Oral Res. 2018;32:e37. doi: 10.1590/1807-3107bor-2018.vol32.0037. Epub 2018 May 3. PMID 29723336
- [Background] Arheiam A, ELTantawi M, ELkadiki N, Elhashani A, Baker SR. Cross-cultural adaptation of the Arabic version of the DHEQ-15. Int J Dent Hyg. 2022 Aug;20(3):527-533. doi: 10.1111/idh.12579. Epub 2022 Jan 28. PMID 35020277
- [Background] Tubert-Jeannin S, Riordan PJ, Morel-Papernot A, Porcheray S, Saby-Collet S. Validation of an oral health quality of life index (GOHAI) in France. Community Dent Oral Epidemiol. 2003 Aug;31(4):275-84. doi: 10.1034/j.1600-0528.2003.t01-1-00006.x. PMID 12846850
- [Background] Allison P, Locker D, Jokovic A, Slade G. A cross-cultural study of oral health values. J Dent Res. 1999 Feb;78(2):643-9. doi: 10.1177/00220345990780020301. PMID 10029462
- [Background] Idon PI, Sotunde OA, Ogundare TO. Beyond the Relief of Pain: Dentin Hypersensitivity and Oral Health-Related Quality of Life. Front Dent. 2019 Sep-Oct;16(5):325-334. doi: 10.18502/fid.v16i5.2272. Epub 2019 Oct 15. PMID 32123872
- [Background] Hirsiger C, Schmidlin PR, Michaelis M, Hirsch C, Attin T, Heumann C, Domejean S, Gernhardt CR. Efficacy of 8% arginine on dentin hypersensitivity: A multicenter clinical trial in 273 patients over 24 weeks. J Dent. 2019 Apr;83:1-6. doi: 10.1016/j.jdent.2019.01.002. Epub 2019 Jan 30. PMID 30710652
- [Background] Terwee CB, Bot SD, de Boer MR, van der Windt DA, Knol DL, Dekker J, Bouter LM, de Vet HC. Quality criteria were proposed for measurement properties of health status questionnaires. J Clin Epidemiol. 2007 Jan;60(1):34-42. doi: 10.1016/j.jclinepi.2006.03.012. Epub 2006 Aug 24. PMID 17161752

DOCUMENTS (1):
  • Study Protocol (2024-06-10): https://cdn.clinicaltrials.gov/large-docs/00/NCT06466200/Prot_000.pdf